CLINICAL TRIAL: NCT04678843
Title: Adapting and Adopting Highly Specialized Pediatric Eating Disorder Treatment to Virtual Care: Implementation Research for the COVID-19 Context and Beyond
Acronym: vFBT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jennifer Couturier (Other)
Responsible Party: Sponsor-Investigator, Jennifer Couturier, Principal Investigator, McMaster University
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12722
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; youth; adolescents; eating disorders; family-based treatment
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: We study a blended implementation approach for Family-Based Treatment delivered via videoconferencing (FBT-V)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Family-Based Treatment (Experimental): Family-based treatment is the gold standard treatment for youth and adolescents with anorexia nervosa. A therapist works with the family to help parents take charge of the process of re-feeding their child, and with progress this control is gradually given back to the youth/adolescent. Other developmental issues are discussed in order to help the youth/adolescent get back to normal development.
  Interventions: Behavioral: Virtual Family-Based Treatment

INTERVENTIONS:
Behavioral: Virtual Family-Based Treatment — Treatment involving the youth/adolescent who has been diagnosed with anorexia nervosa and their family, delivered virtually via videoconferencing.

SUMMARY:
The COVID-19 pandemic has had detrimental effects on mental health. Individuals with eating disorders (EDs) are no exception, exhibiting increased symptoms and exacerbated feelings of isolation and anxiety. Across Canada, in-person outpatient services have been quickly replaced with virtual care, yet practitioners and patients have noted substantial challenges in adapting ED-related care virtually. Given the success of our previous research on Family-Based Treatment (FBT) for EDs, as well as the rapid transition to virtual care during COVID-19, there is an urgent need to adapt FBT to virtual formats and adopt it in the ED network. Using a multi-site case study with a mixed method pre/post design, this study aims to examine the implementation of virtual FBT (vFBT) as well as its impact within six ED programs in Ontario, building on the investigator's previous work, and further developing capacity in the system. The investigator will develop implementation teams at each site and provide a virtual training workshop on vFBT, with ongoing consultation during initial implementation. The investigator proposes to examine implementation success by studying fidelity to vFBT, as well as team and patient/family experience with virtual care, and patient outcomes. These findings for virtual care will not only be important in the COVID-19 context but are also vital in the North, where access to specialized services is extremely limited.

ELIGIBILITY:
Inclusion Criteria:

* Youth must be under 18 years of age in order to participate
* Youth must have a diagnosis of Anorexia Nervosa in order to participate
* Must have the capacity to write, speak, and understand English
* Must have access to a computer and the internet.

Exclusion Criteria:

* Individuals 18 years of age and older are unable to participate
* Youth without a diagnosis of Anorexia Nervosa are unable to participate
* Individuals who cannot write, speak and understand English are unable to participate
* Individuals who do not have access to a computer and the internet are unable to participate

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Key components of FBT | Completed after session 4 of treatment, approximately 4 months
  Measured by a self-report questionnaire entitled Key Measure of Therapist Behaviours and Self-Efficacy in FBT (an indicator of therapist adherence to the key components of standard FBT within the vFBT model)
Fidelity | Completed after the session 4 of treatment, approximately 4 months
  Fidelity to vFBT, measured by FBT fidelity ratings of the first four sessions of vFBT using the FBT Fidelity and Adherence Check (experts in FBT fidelity rating will rate the recordings).

SECONDARY OUTCOMES:
Qualitative experience of participants | Completed after session 4 of treatment, approximately 4 months
  Experiences of the therapists, medical practitioners, administrators, and families in vFBT, qualitatively measured during semi-structured focus groups
Change in Weight | At baseline before treatment, and at 1 week, 2 weeks, 3 weeks, and 4 weeks.
  Weight will be measured in kilograms.
Change in Number of Binge/Purge Episodes | At baseline before treatment, and at 1 week, 2 weeks, 3 weeks, and 4 weeks.
  The number of binge/purge episodes each week will be recorded by patients/their families.
Therapists' Change in Readiness | At baseline, after training (approx. 1 month), and after 4 sessions of treatment (approx. 4 months)
  The Brief Individual Readiness to Change Scale will indicate how ready therapists feel they are to change. Higher scores indicate greater readiness to use research-based direct service techniques. Minimum score is 0, maximum score is 20.
Therapists' Change in Attitudes about Evidence Based Practice | At baseline, after training (approx. 1 month), and after 4 sessions of treatment (approx. 4 months)
  Their attitudes about evidence-based practice will be assessed using the Evidence Based Practice Attitudes Scale (EBPAS). The subscales include requirements, appeal, openness and divergence. The score for each subscale is created by computing a mean score for the items that load on a given subscale. Minimum score for each subscale is 0, maximum score for each subscale is 4.
Therapists' Change in Confidence related to the Intervention | At baseline, after training (approx. 1 month), and after 4 sessions of treatment (approx. 4 months)
  Their confidence related to the intervention will be assessed by administering an adapted version of the Perceived Attributes of the Principles of Effectiveness Scale (MPAS). Higher scores are indicative of more favorable perception for FBT content. The minimum score is 18, the maximum score is 90.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Couturier, MD MSc, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - St. Joseph's Care Group, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - CMHA Waterloo Wellington, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Couturier J, Pellegrini D, Grennan L, Nicula M, Miller C, Agar P, Webb C, Anderson K, Barwick M, Dimitropoulos G, Findlay S, Kimber M, McVey G, Lock J. Multidisciplinary implementation of family-based treatment delivered by videoconferencing (FBT-V) for adolescent anorexia nervosa during the COVID-19 pandemic. Transl Behav Med. 2023 Feb 28;13(2):85-97. doi: 10.1093/tbm/ibac086. PMID 36327378
- [Derived] Couturier J, Pellegrini D, Grennan L, Nicula M, Miller C, Agar P, Webb C, Anderson K, Barwick M, Dimitropoulos G, Findlay S, Kimber M, McVey G, Paularinne R, Nelson A, DeGagne K, Bourret K, Restall S, Rosner J, Hewitt-McVicker K, Pereira J, McLeod M, Shipley C, Miller S, Boachie A, Engelberg M, Martin S, Holmes-Haronitis J, Lock J. A qualitative evaluation of team and family perceptions of family-based treatment delivered by videoconferencing (FBT-V) for adolescent Anorexia Nervosa during the COVID-19 pandemic. J Eat Disord. 2022 Jul 26;10(1):111. doi: 10.1186/s40337-022-00631-9. PMID 35883167
- [Derived] Couturier J, Pellegrini D, Miller C, Agar P, Webb C, Anderson K, Barwick M, Dimitropoulos G, Findlay S, Kimber M, McVey G, Lock J. Adapting and adopting highly specialized pediatric eating disorder treatment to virtual care: a protocol for an implementation study in the COVID-19 context. Implement Sci Commun. 2021 Apr 8;2(1):38. doi: 10.1186/s43058-021-00143-8. PMID 33832543